CLINICAL TRIAL: NCT02230293
Title: Assistance Multidisciplinary in Hypertensive Patient: Randomized Clinical Trial
Acronym: MULTIHAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Silvia Goldmeier, Doctor, Instituto de Cardiologia do Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UP 3927-06
Record Dates: First submitted 2014-08-06; First posted 2014-09-03 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Hypertension
Keywords: ambulatory care,; hypertension,; health personnel,; clinical trial
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Group (Active Comparator): Conventional treatment and follow up
  Interventions: Other: Conventional treatment and follow up
- Multidisciplinary Group (Experimental): Multidisciplinary assistance
  Interventions: Other: Multidisciplinary assistance

INTERVENTIONS:
Other: Multidisciplinary assistance — Multidisciplinary group assistance was effected every two months by all professionals (physician, nurse, dietitian, physiotherapist and psychologist) and consisted in orientations and mechanisms to medication and non-pharmacological adherence (lifestyle changes).
  Arms: Multidisciplinary Group
Other: Conventional treatment and follow up — Assistance was effected by physician and nurse and consisted about adapting to the drug
  Arms: Conventional Group

SUMMARY:
The purpose of this study is to determine if multidisciplinary care improves the health condition of hypertensives.

DETAILED DESCRIPTION:
A multidisciplinary approach in managing hypertensive patients has shown benefits in reducing blood pressure and risk factors for hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years of age
* Diagnosis of hypertension

Exclusion Criteria:

* Secondary hypertension
* Hypertensive patients with congenital cardiopathy
* Surgical patients
* Proven myocardial infarction

Ages: 41 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2008-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Systolic and Diastolic Blood pressure | Measured at the first appointment and 1 year later

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Goldmeier, Dr, Study Chair — Instituto de Cardiologia do Rio Grande do Sul
Locations (1):
- Instituto de Cardiologia do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil